CLINICAL TRIAL: NCT04428164
Title: Enhancing Patient Experience of Pain and Sleep Through Non-Pharmacological Strategies
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 075.NUR.2019.A
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Comfort

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalized patients: Any patient admitted to the study units (MDMC: 10ST; MCMC: A6; MMMC: A3; MRMC: 3Medical ) that do not have any of the exclusion criteria
  Interventions: Other: The Richards-Campbell Sleep Questionnaire (R-CSQ); Other: Revised American Pain Society Outcome Questionnaire (APS-POQ-R)

INTERVENTIONS:
Other: The Richards-Campbell Sleep Questionnaire (R-CSQ) — Tool developed to assess patient satisfaction and comfort in the hospital setting.
  The R-CSQ is a scale used to measure different aspects of sleep quality. This scale allows the patient to rate their quality and amount of sleep on a scale of 0-100. The R-CSQ allows the patient to rate six different components of their sleep, including sleep depth, sleep latency, awakenings, returning to sleep, sleep quality, and noise.
Other: Revised American Pain Society Outcome Questionnaire (APS-POQ-R) — The APS-POQ-R can be utilized to measure perceived levels of pain in patients. The APS-POQ-R scale is a validated scale that is used in the hospital setting with reliable and consistent results. This scale measures five aspects of a patient's perception and experiences with pain and a sixth aspect including nonpharmacological interventions.

SUMMARY:
Comfort can be a physical sensation, a psychological state, or both simultaneously . Patient comfort in an inpatient setting is a subjective state that varies from each individual based on different factors and situations. The Richards-Campbell Sleep Questionnaire (R-CSQ) and the Revised American Pain Society Outcome Questionnaire (APS-POQ-R) are tools that have been developed to assess patient satisfaction and comfort in the hospital setting. The R-CSQ is a scale used to measure different aspects of sleep quality. This scale allows the patient to rate their quality and amount of sleep on a scale of 0-100. The R-CSQ allows the patient to rate six different components of their sleep, including sleep depth, sleep latency, awakenings, returning to sleep, sleep quality, and noise. The APS-POQ-R can be utilized to measure perceived levels of pain in patients. The APS-POQ-R scale is a validated scale that is used in the hospital setting with reliable and consistent results. This scale measures five aspects of a patient's perception and experiences with pain and a sixth aspect including nonpharmacological interventions.

We propose that if patients implement interventions that promote sleep and decrease pain, comfort will be improved.

DETAILED DESCRIPTION:
Aim(s)/Objective(s)

* Improve patient sleep during their hospital stay.
* Determine patient self-reported pain assessment using non-pharmacologic strategies.
* Determine if the "patient toolkit" improves patient experience of pain and sleep.

Hypothesis 1. Primary Hypothesis Patients' experience of pain and sleep will improve with the implementation of interventions from our "patient toolkit".

.2. Secondary Hypothesis Patients will report an increase in sleep and a decrease in pain after use of the interventions provided in the "patient toolkit".

3. Tertiary Hypothesis Patients will report satisfaction with results gained through implementation of our "patient toolkit".

STUDY DESIGN

* 60 to 80 medical surgical patients per campus (MCMC, MDMC, MMMC, MRMC) will be recruited to participate (total: 240 to 320 patients) Only adult medical surgical patients over the age 20 will be recruited.
* Quasi-experimental, pre-/post-test, repeated measures interventional study
* Length of patients hospital stay will determine length of intervention used; average estimate is a four-day length of stay
* Give pre-assessment the morning after first night of admission (Day 2)
* Participants will receive a toolkit upon informed consent completion that will include intervention strategies (eye mask; ear plugs; puzzle book; adult coloring book; colored pencils; aromatherapy patches; herbal tea bags) and data collection booklet for pre-survey, daily survey, and post-survey
* Data will be collected over 6 to 10 weeks to achieve desired number of participants
* Anticipated completion of study will be December 2021

ELIGIBILITY:
Inclusion Criteria:

Hospitals eligible to participate will meet the following criteria:

* Part of the MHS (MCMC, MDMC, MMMC, MRMC)
* The hospital has at least one clinical site/sub-investigator on-staff
* Hospital has 150 or more inpatient beds

Patients eligible to participate will meet the following criteria:

* Any patient admitted to the study units (MDMC: 10ST; MCMC: A6; MMMC: A3; MRMC: 3Medical ) that do not have any of the exclusion criteria described below
* Age: 20+ y/o
* Must be able to speak/read/write/understand English
* Willing to utilize study interventions and complete survey booklet

Exclusion Criteria:

Hospitals outside of MHS will be excluded.

Patients will be excluded for the following reasons:

* Patients admitted for surgical procedure
* Change in clinical status and deterioration requiring higher level care
* Altered mental status
* Any history of dementia and/or Alzheimer's
* Disoriented/confused
* Patients suffering with chronic pain
* Patients on patient-controlled analgesia
* Observation status patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 to 80 medical surgical patients per campus (MCMC, MDMC, MMMC, MRMC) will be recruited to participate (total: 240 to 320 patients) Only adult medical surgical patients over the age 20 will be recruited.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Perception of Pain | From January 2021 until December 2021
  The Revised American Pain Society Patient Outcome Questionnaire will measure patient perception of pain. This scale measures five aspects of patient's perception and experiences with pain and a sixth aspect including nonpharmacological interventions. The scale goes from (0) - No pain to (10) - Worst Pain Possible

SECONDARY OUTCOMES:
Sleep Quality | From January 2021 until December 2021
  The Richards-Campbell Sleep Questionnaire (R-CSQ) will measure different aspects of sleep quality. The R-CSQ allows the patient to rate six different components of their sleep, including sleep depth, sleep latency, awakenings, returning to sleep, sleep quality, and noise.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sweatt, MSN, RN, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No